CLINICAL TRIAL: NCT07302516
Title: A Multi-center, Randomised, Double Blind, Active Controlled Phase III Trial to Compare the Efficacy and Safety of QL2302 With Tezspire® in Adults With Uncontrolled Severe Asthma
Brief Title: Compare the Efficacy and Safety of QL2302 Versus Tezspire® in Severe Asthma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL2302-301
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2302 (Experimental)
  Interventions: Biological: tezepelumab (Arm1&Arm2)
- Tezspire® (Active Comparator)
  Interventions: Biological: tezepelumab (Arm1&Arm2)

INTERVENTIONS:
Biological: tezepelumab (Arm1&Arm2) — 210mg Q4W (Arm1&Arm2)

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of QL2302 and Tezspire® in patients with uncontrolled severe asthma. The main questions it aims to answer are:

* if the efficacy of QL2302 and Tezspire® are similar
* if the safety of QL2302 and Tezspire® are similar

Participants will be randomised to QL2302 or Tezspire® group and asked to receive one injection of QL2302 or Tezspire® subcutaneously every four weeks till Week 48, which means participants will receive a total of 13 injections. And be observed for another 12 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 year of age
2. Body weight ≥40 kg
3. Diagnosed with asthma ≥12 months
4. Received a total daily dose of medium/high dose of ICS for more than 3 months steadily
5. At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.
6. Morning pre-BD FEV1 <80% but ≥35% predicted normal
7. Evidence of asthma as documented by reversibility test or change of PEF.
8. Documented history of at least 1 asthma exacerbation events within 12 months.
9. ACQ-5 score ≥1.5 at screening and on day of randomization

Exclusion Criteria:

1. Pulmonary disease other than asthma.
2. History of cancer within 5 years except those cured.
3. History of a clinically significant infection within 4 weeks.
4. Current smokers or participants with smoking history ≥10 pack-yrs.
5. History of chronic alcohol or drug abuse within 12 months.
6. Positive Hepatitis B, C or HIV infection.
7. Pregnant or breastfeeding.
8. History of anaphylaxis following any biologic therapy.
9. Participant received tezepelumab or other TSLP antibody priorly.
10. Participant received bronchial thermoplasty within 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint ： | 52 weeks
  Annualized Asthma Exacerbation Rate (AAER)